CLINICAL TRIAL: NCT07080619
Title: A Phase IIa Clinical Study to Assess the Efficacy and Safety of SC-101 in Patients With Advanced Malignant Tumors Positive for NECTIN4 Gene Amplification
Brief Title: SC-101 in Subjects With Advanced NECTIN4-Amplified Cancers
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin ConjuStar Biologics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-101-201
Record Dates: First submitted 2025-07-07; First posted 2025-07-23 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: TNBC - Triple-Negative Breast Cancer; HR+ Breast Cancer
Keywords: SC-101
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TNBC, HR+HER2- BC, and other tumors (Experimental): Receive 7.5 mg/m² of SC-101 intravenously once weekly (QW).
  Interventions: Drug: SC-101

INTERVENTIONS:
Drug: SC-101 — Receive 7.5 mg/m² of SC-101 intravenously once weekly (QW).

SUMMARY:
This study is an open-label, multicenter Phase IIa trial to evaluate the efficacy and safety of SC-101 monotherapy in patients with locally advanced or metastatic malignant tumors who are positive for NECTIN4 gene amplification.

DETAILED DESCRIPTION:
The study will include multiple cohorts: triple-negative breast cancer (TNBC), HR-positive HER2-negative breast cancer, and other solid tumors.

Participants will receive SC-101 at a dose of 7.5 mg/m² once weekly, with treatment cycles lasting 28 days. The study aims to assess tumor response and safety until disease progression or other reasons for treatment discontinuation.

Eligibility requires patients to have locally advanced or metastatic tumors that have either relapsed after standard treatment, are resistant to treatment, or are not amenable to standard treatment. NECTIN4 gene amplification must be confirmed via tumor tissue testing.

Imaging assessments will be conducted every 8 weeks to evaluate tumor response. Safety follow-up will be performed 30 days after the last dose, with additional survival follow-ups every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 75 years (inclusive), regardless of gender.

ECOG performance status of 0-1.

Expected survival of more than 3 months, as assessed by the investigator.

Fertile participants must agree to use contraception.

Able to understand the trial requirements and willing and able to comply with the trial and follow-up procedures.

Adequate bone marrow and organ function.

NECTIN-4 gene amplification positive.

Exclusion Criteria:

Unstable central nervous system tumors.

Adverse reactions from previous anticancer treatments have not recovered to a CTCAE 5.0 grade ≤1.

A history of severe cardiovascular or cerebrovascular disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
cORR | Baseline (Day -28 to Day -1); tumor response will be evaluated every 8 weeks (±7 days) from the first dose of study treatment to the data cut-off date, up to 24 months.
  Investigator-assessed confirmed objective response rate

IPD SHARING:
Plan to Share IPD: Undecided
The data sharing plan has not been determined yet and will be further clarified after the study begins.